CLINICAL TRIAL: NCT02889237
Title: Assessment of Fracture Healing by High-resolution Peripheral Quantitative Computed Tomography (HR-pQCT) and Bone Strength Analysis in Standard Care and After Immediate Administration of Calcium and Vitamin D Supplementation
Brief Title: Fracture Healing Assessed by HR-pQCT After Administration of Calcium and Vitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VieCuri Medical Centre (Other)
Responsible Party: Principal Investigator, Joop P.W. van den Bergh, Prof. dr. J.P.W. van den Bergh, Endocrinologist, VieCuri Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NL46035.072.13
Record Dates: First submitted 2014-09-26; First posted 2016-09-05 (Estimated); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Bone Fracture
Keywords: Fracture healing; Calcium supplementation; Vitamin D supplementation; HR-pQCT
MeSH Terms: conditions — Fractures, Bone | interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Standard care (No Intervention): Start of calcium and vitamin D3 supplementation according to standard care, i.e. 12 weeks after fracture.
- Calcium (Active Comparator): Immediate administration of daily calcium supplementation (1000 mg calcium)
  Interventions: Dietary Supplement: Calcium
- Calcium and low dose vitamin D (Active Comparator): Immediate administration of daily calcium + low dose vitamin D supplementation (1000 mg calcium + 880 IU vitamin D).
  Interventions: Dietary Supplement: Calcium + low dose vitamin D
- Calcium and high dose vitamin D (Active Comparator): Immediate administration of daily calcium + high dose vitamin D supplementation (1000 mg calcium + 1760 IU vitamin D)
  Interventions: Dietary Supplement: Calcium + high dose vitamin D
- Already on treatment with Calcium or vitamin D (No Intervention): Patients who are already treated with Calcium or Vitamin D.

INTERVENTIONS:
Dietary Supplement: Calcium — Immediate administration of daily calcium supplementation for 12 weeks
  Other Names: Cacit effervescent tablet '1000'
  Arms: Calcium
Dietary Supplement: Calcium + low dose vitamin D — Immediate administration of daily calcium and low dose vitamin D (1 sachet CaD 1000/880) supplementation for 12 weeks
  Other Names: CaD® sachet 1000/880
  Arms: Calcium and low dose vitamin D
Dietary Supplement: Calcium + high dose vitamin D — Immediate administration of daily calcium and high dose vitamin D (2 sachets CaD 500/880) supplementation for 12 weeks
  Other Names: CaD® sachets 500/880
  Arms: Calcium and high dose vitamin D

SUMMARY:
This study is designed as a single-blind RCT in 80 postmenopausal women to compare the effect of immediate administration of daily calcium supplementation (1000 mg calcium) or two daily dosages of calcium + vitamin D (1000 mg calcium + 880 IU vitamin D or 1000 mg calcium + 1760 IU vitamin D) to standard care (administration of vitamin D3 12 weeks after fracture) in terms of calculated bone strength based on analysis of cortical and trabecular bone parameters using HR-pQCT, fracture healing and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women older than 50 years who present themselves in clinic with a distal radius fracture due to a trauma.
* Patients with a stable distal radius fracture treated by cast immobilization.
* Patients who understand the conditions of the study and are willing and able to comply with the scheduled biochemical and radiographic evaluations and the prescribed rehabilitation.
* Patients who signed the Ethics Committee approved specific Informed Consent Form prior to inclusion.

Exclusion Criteria:

* Patients who underwent surgery of the wrist or radius on a previous occasion on the same side or who need surgery this time.
* Patients with active or suspected infection such as pneumonia or complicated urinary tract infection in the last 3 months.
* Patients with malignancy or a pathological fracture in the last 12 months.
* Patients with a neuromuscular or neurosensory deficit, e.g. Parkinson's disease, which would limit the ability to assess the performance during the healing period.
* Patients with known systemic or metabolic disorders leading to progressive bone deterioration, such as: hyperthyroidism, hyperparathyroidism, chronic kidney disease with eGFR<30 ml/min, sarcoidosis, hypercalcemia,
* Patients with an active inflammatory disease during the last year such as rheumatoid arthritis, systemic lupus erythematous, inflammatory bowel disease, e.g. Crohn's disease and ulcerative colitis.
* The use of glucocorticoids during the last 12 months.
* Patients with an allergy to calcium, calcium carbonate, cholecalciferol, aspartame, citric-acid, lactose, dimethicone, methylcellulose, sorbic acid, macrogole, polyvidone, mannitol, orange flavour, natriumsaccharine, starch or sucrose.
* Patients, who as judged by the principal Investigator, are mentally incompetent or are unlikely to be compliant with the follow-up evaluation schedule.
* Patients with other severe concurrent joint involvements that can affect their outcome.
* Patients who are already selected for another trial concerning distal radius fractures.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Bone strength | 1 year
  Bone strength parameters will be assessed by HRpQCT

SECONDARY OUTCOMES:
Fracture healing | 1 year
Functional outcome assessed by PRWE | 1 year
  Functional outcome is assessed using Patient-Related Wrist Examination (PRWE) questionnaire
Functional outcome assessed by QuickDASH | 1 year
  Functional outcome is assessed using QuickDASH questionnaires
Functional outcome assessed using VAS for pain score | 1 year
  Functional outcome is assessed using VAS for pain score on Visual Analogue Scale (VAS)
Functional outcome assessed using range of motion | 1 year
  Functional outcome is assessed by measuremt of range of motion of the fractured wrist

CONTACTS AND LOCATIONS:
Overall Officials: J PW van den Bergh, MD, PhD, Principal Investigator — VieCuri Medical Centre
Locations (1):
- VieCuri Medical Centre, Venlo, Limburg, Netherlands